CLINICAL TRIAL: NCT00457951
Title: An Open-Label Phase Followed by a Randomized, Double-Blind, Placebo-Controlled Phase in a Study Designed to Evaluate Intravenous 2-O, 3-O Desulfated Heparin (ODSH) in Subjects With Exacerbations of Chronic Obstructive Pulmonary Disease
Brief Title: A Study Designed to Evaluate ODSH in Subjects With Exacerbations of COPD
Acronym: COPD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim analysis: safety without efficacy ODSH in patients with acute COPD.
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PGX-ODSH-2006
Record Dates: First submitted 2007-04-06; First posted 2007-04-09 (Estimated); Results first posted 2016-12-16 (Estimated); Last update posted 2021-12-02 (Actual); Status verified 2016-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; COPD; Heparin; ODSH; Exacerbations of COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Open Label (Experimental): Initial six subjects treated with ODSH open-label to confirm safety in subjects with an acute exacerbation of COPD; six additional patients will be enrolled following safety review.
  Interventions: Drug: Open-Label
- 0.9% Sodium Chloride (Placebo Comparator): Placebo Comparator: Placebo-Control Arm 0.9% Sodium Chloride Solution bolus; dose of 0.375mg/kg/hr over 96 hours.
  Interventions: Drug: Placebo Comparator: Placebo-Control Arm 0.9% Sodium Chloride
- Randomized, Blinded, ODSH Arm (Active Comparator): Subjects will receive standard of care treatment. ODSH is administered in bolus doses estimated to inhibit inflammatory mediators randomized 1:1 to ODSH 8mg/kg or placebo. The continuous infusion dose will be 0.375 mg/kg/hr over 96 hours.
  Interventions: Drug: ODSH

INTERVENTIONS:
Drug: Open-Label — ODSH administered open-label
  Other Names: PGX-100
  Arms: Open Label
Drug: Placebo Comparator: Placebo-Control Arm 0.9% Sodium Chloride — Placebo-Control Arm: Bolus infusion followed by a 96 hour continuous infusion of 0.9%Sodium Chloride
  Other Names: 0.9% Sodium Chloride Solution Placebo-Control Arm
  Arms: 0.9% Sodium Chloride
Drug: ODSH — Randomized, Blinded, ODSH Arm
  Other Names: PGX-100
  Arms: Randomized, Blinded, ODSH Arm

SUMMARY:
The purpose of this study is to determine whether ODSH, when added to conventional treatment, is more effective in treating COPD exacerbations than conventional therapy alone.

DETAILED DESCRIPTION:
The management of acute exacerbations of COPD today is qualitatively the same as it was 40 years ago: bronchodilators, corticosteroids, and antibiotics. Because of the prominent pathophysiological role of neutrophils in exacerbations of COPD, neutrophils and their toxic oxidants and proteases represent therapeutic targets which are currently unchallenged in the treatment of this aspect of the disease. Ideally, to disrupt neutrophilic airway inflammation, one would both block neutrophilic influx from the vascular space into the airway, as well as neutralize or inactivate prominent neutrophilic toxins such as the proteases HLE and cathepsin G.

Heparin is a sulfated mucopolysaccharide that slows blood clot formation by inhibiting the reactions that lead to formation of fibrin clots. Physicians use heparin to prevent blood clot formation during open-heart surgery, bypass surgery and dialysis. Heparin also prevents previously formed clots from becoming larger and causing more serious problems. Heparin has other biological properties, most notably anti-inflammatory activity. At doses required to be therapeutically beneficial as an anti-inflammatory, heparin can cause severe, potentially life-threatening hemorrhage. ParinGenix has chemically modified heparin to retain the anti-inflammatory activity while reducing anti-coagulant properties.

Heparin has long been known to be a potent inhibitor, both in vitro and in vivo, of the cationic neutrophil proteases HLE and cathepsin G. However, heparin also has numerous other important anti-inflammatory effects. P-selectin is the primary endothelial attachment molecule mediating neutrophil rolling along the vessel wall. At concentrations close to those achieved in plasma near the high range of therapeutic anticoagulation, heparin inhibits P-selectin and P-selectin mediated interaction of leukocytes with endothelium. Heparin also blocks the leukocyte integrin Mac-1 (CD11b/CD18) and Mac-1-dependent leukocyte adherence to endothelial ICAM. These combined effects on rolling, integrin-dependent attachment and perhaps other aspects of cellular passage through the basement membrane prevent neutrophil accumulation in areas of inflammation. As an example, when given in much higher concentrations than those appropriate for therapeutic anticoagulation, heparin efficiently blocks neutrophilic influx into ischemic reperfused myocardium and brain reducing the size of both myocardial infarction and ischemic stroke. Thus, heparin and heparin analogues may have the potential to also reduce inflammatory influx of neutrophils into the airway during exacerbations of COPD.

All subjects will receive standard of care treatment, including corticosteroids, beta-2 agonists, and antibiotics as well as ODSH or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients (40 years of age or older) with an established diagnosis of COPD based upon medical history who are being admitted to the hospital to treat an exacerbation of COPD;
2. Normal prothrombin time and activated partial thromboplastin time; Platelet count; hemoglobin and hematocrit

Exclusion Criteria:

1. Certain diseases such as:

   * asthma;
   * left heart failure or pulmonary embolism;
   * lung cancer;
   * pneumonia
   * liver or kidney disease
   * blood clotting disorder
   * Positive HIV or hepatitis tests
   * GI bleeding, physical trauma with bleeding, any disease with bleeding within 60 days of study entry
2. Certain medications such as:

   * Plavix®
   * Warfarin
   * Heparin therapy
   * Certain antibiotics
3. Exacerbations that are too severe (requiring intubation and mechanical ventilation)
4. Women of child-bearing potential, pregnancy or breast-feeding
5. Unable or unwilling to provide informed consent and follow study procedures.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2007-04; Primary Completion 2009-08 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Welte, MD, Principal Investigator — Hannover Medical School
Locations (38):
- United States (10):
  - Pulmonary Consultants & Primary Care, Orange, California
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Louisiana State University Health Sciences Center in Shreveport, Shreveport, Louisiana
  - Washington Universtiy School of Medicine, St Louis, Missouri
  - The Oregon Clinic, Portland, Oregon
  - Temple University of the Commonwealth of Higher Education, Philadelphia, Pennsylvania
  - Methodist Hospital, Houston, Texas
  - Michael E. DeBakey VA Medical Center, Houston, Texas
  - University of Texas Health Care Center at Tyler, Tyler, Texas
  - Western Washington Medical Group, Everett, Washington
- Belgium (3):
  - University Hospital Gasthuisberg, Leuven
  - CHU Liege Domain Universitaire du Sart Tilman, Liège
  - Cliniques Universiaries U.C.L. de Mont-Gondinne, Yvior
- Canada (9):
  - University of Alberta Hospital, Edmonton, Alberta
  - Kelowna General Hospital, Kelowna, British Columbia
  - Vancouver Coastal Health, Vancouver, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - QE II Health Sciences Centre, Halifax, Nova Scotia
  - Credit Valley Hospital,, Mississauga, Ontario
  - The Ottawa Hospital, Civic Campus, Ottawa, Ontario
  - University of Toronto, Toronto, Ontario
  - Laval Hospital, Québec, Quebec
- Germany (5):
  - Klinik Schillerhohe, Gerlingen
  - Pneumologisches Forschungsinstitut GmbH, Großhansdorf
  - Medizinsche Hochschule, Hanover
  - Uniklinikum Mainz, Mainz
  - Klinikum der LMU Innenstadt, München
- Poland (11):
  - Wojewodzki Szpital Specjalistyczny im. Najswietszej Marii Panny, Częstochowa
  - Samodzielny Publiczny Szpital Kliniczny SUM w Katowicach, Katowice
  - Krakowski Szpital Specjalistyczny im. Jana Pawla II, Krakow
  - Samodzielny Publiczny ZOZ, Uniwersytecki Szpital Liniczny nr 1 im Norberta Barlickiego, Lodz
  - Wojewodzki Szpital Specjalistyczny im. Stefana Kardynala Wyszynskiego, Samodzielny Publiczny Zespol Opieki Zdrowotnej, Lublin
  - Samodzielny Publiczny Szpital Klinczny nr 4 W Lublinie, Lublin
  - Zespol Opieki Zdrowotnej w Olawie, Oława
  - Wieklopolskie Centrum Chorob Pluc i Gruzlicy, Poznan
  - I Klinika Chorob Plus, Instyut Gruzlicy i Chorob Pluc, Warsaw
  - Miedzyleski Szpital Specjalistyczny w Warszawie, Warsaw
  - Akademicki Szpital Kliniczny im. Jana Mikulicza-Radeckiego, Wroclaw

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Label: Open Label
  The original protocol called for 304 subjects with exacerbation of COPD to be enrolled into the study. Thirteen patients with exacerbation of COPD were enrolled in the initial open label portion of the study. Of these thirteen subjects, the initial seven subjects were treated with an IV bolus of ODSH at 8 mg/kg followed by a continuous infusion of ODSH at 0.5 mg/kg/hr for 72 hours.
  After an ad hoc safety committee assessed the safety of the data from the first seven subjects, six more subjects were treated concomitantly treated with ODSH and enoxaparin, a low molecular weight heparin commonly used for seriously ill hospitalized patients as DVT prophylaxis.
- Placebo Comparator: 0.9% Sodium Chloride: Double-blind randomized phase: Normal Saline infusion: Bolus infusion followed by a 4 day continuous infusion of placebo.
- ODSH Treatment Group: Double-blind randomized phase: The subjects receiving ODSH in the randomized portion of the study received 0.375 mg/kg/hr continuous IV infusion of ODSH for 96 hours.
Period: Overall Study
Arm/Group | Open Label | Placebo Comparator: 0.9% Sodium Chloride | ODSH Treatment Group
Started (In the double-blind phase, 145 subjects consented and 138 met criteria and were randomized.) | 13 | 66 | 72
Completed | 13 | 50 | 60
Not Completed | 0 | 16 | 12

BASELINE CHARACTERISTICS:
Population: Open-Label followed by multi-center, randomized, double-blind, placebo-controlled trial in hospitalized subjects with exacerbations of COPD. In the double-blind phase, 145 subjects consented and 138 met criteria and were randomized.
Groups:
- Open-Label: Open-Label ODSH
- Placebo Comparator: Placebo-Control: 0.9% Sodium Chloride: Placebo Comparator: Placebo-Control: 0.9% Sodium Chloride Administered as bolus; then continuous administration over 96 hours in hospitalized subjects with exacerbations of COPD
- ODSH Treatment Group: ODSH Treatment Group Administered as bolus; then continuous administration over 96 hours in hospitalized subjects with exacerbations of COPD
- Total: Total of all reporting groups
Arm/Group | Open-Label | Placebo Comparator: Placebo-Control: 0.9% Sodium Chloride | ODSH Treatment Group | Total
Number analyzed (Participants) | 13 | 66 | 72 | 151
Age, Customized [Mean (Standard Deviation); unit: years] | 63.8 (15) | 68.5 (10.24) | 67.2 (9.53) | 66.5 (10.43)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 9 | 25 | 23 | 57
  Male | 4 | 41 | 49 | 94
Region of Enrollment [Number; unit: participants]
  United States | 13 | 66 | 72 | 151

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment Failure
Description: The primary outcome of the study is "Treatment Failure" as defined by Failure to discharge from hospital based on GOLD (Global Strategy for the Diagnosis, Management, and Prevention of Chronic Obstructive Pulmonary Disease) criteria or relapse after DC from hospital.
Time Frame: Time to hospital discharge and 21 days post-treatment, up to 31 days
Population: Of the 138 subjects randomized, 132 were analyzed in the intent-to-treat population. Of the 6 excluded from the intent-to-treat population, 4 did not receive study drug and 2 lacked information for assessment.
Measure: Number (95% Confidence Interval); unit: percentage of failures
Arm/Group | 0.9% Sodium Chloride | Randomized, Blinded, ODSH Arm
Number analyzed (Participants) | 64 | 68
percentage of failures | 24.6 [14 to 43] | 32.4 [21 to 42]

ADVERSE EVENTS:
Time Frame: D1 to D90
Description: Of the 145 subjects consented in the randomized phase, 138 were randomized. Of the 138 randomized subjects, 134 were included in the safety population; 4 of the 138 randomized subjects did not receive study medication.
Groups:
- Placebo Comparator: 0.9% Sodium Chloride: Placebo Comparator: Placebo-Control Arm 0.9% Sodium Chloride Solution bolus; dose of 0.375mg/kg/hr over 96 hours.
  Placebo Comparator: Placebo-Control Arm 0.9% Sodium Chloride: Placebo-Control Arm: Bolus infusion followed by a 96 hour continuous infusion of 0.9%Sodium Chloride
- ODSH Treatment Group: Subjects will receive standard of care treatment. ODSH is administered in bolus doses estimated to inhibit inflammatory mediators randomized 1:1 to ODSH 8mg/kg or placebo. The continuous infusion dose will be 0.375 mg/kg/hr over 96 hours.
  ODSH: Randomized, Blinded, ODSH Arm
Arm/Group | Open Label | Placebo Comparator: 0.9% Sodium Chloride | ODSH Treatment Group
Serious Adverse Events (participants affected / at risk) | 1/13 | 4/65 | 2/69
Other Adverse Events (participants affected / at risk) | 0/13 | 13/65 | 48/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open Label (N=13) | Placebo Comparator: 0.9% Sodium Chloride (N=65) | ODSH Treatment Group (N=69)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Guillain-barre syndrome (Nervous system disorders) | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label (N=13) | Placebo Comparator: 0.9% Sodium Chloride (N=65) | ODSH Treatment Group (N=69)
ALT Increased (Hepatobiliary disorders) | 0 (0) | 7 (8) | 26 (33)
AST Increased (Hepatobiliary disorders) | 0 (0) | 6 (6) | 22 (29)
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 4
Constipation (Gastrointestinal disorders) | 0 | 1 | 4

LIMITATIONS AND CAVEATS:
PGX-ODSH-2006, Ph II in patients with exacerbation of COPD. There were no safety issues. An interim analysis demonstrated lack of efficacy for the primary and secondary endpoints; therefore, Cantex terminated the study on August 11, 2009.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Confidentiality and Non-Disclosure Agreement